CLINICAL TRIAL: NCT05087433
Title: The Effect of Web-based Progressive Relaxation Exercises on Perceived Stress and Anxiety on Nurses Working in a Pandemic Hospital: A Randomized Controlled Trial
Brief Title: Perceived Stress and Anxiety Levels of Nurses
Acronym: stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe Aydınlı (Other)
Responsible Party: Sponsor-Investigator, Ayşe Aydınlı, Research Asistant, RN, MsN, PhD, Suleyman Demirel University
Organization: Suleyman Demirel University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Stress and Anxiety
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Stress; Anxiety
Keywords: Anxiety; Pandemics; Nurse; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention Group (Experimental): Practicing Progressive Relaxation Exercises The training of the Zoom application progressive relaxation exercise for the nurses was done in two sessions for a total of 60 minutes. During the first interview, the definition, purpose, benefits, and application techniques of PRE were explained to the nurses in the intervention group. In the second session, the steps of progressive relaxation exercises were demonstrated by the trainer.
  The trainer performed the PRE exercise online with the nurses. Nurses were asked to perform the PRE application in accordance with the commands in the video recordings. In addition, a guide in which the steps of applying progressive relaxation exercises for each muscle group were written was given to the nurses. It was stated that they should do the application regularly for 25-30 minutes in the morning every day at home for a month.
  Interventions: Other: Progressive Relaxation Exercises
- Control Group (No Intervention): No intervention was applied to the control group during the study. However, after the research was completed, the video of the application of the progressive relaxation exercises to the control group was shared on the WhatsApp group.

INTERVENTIONS:
Other: Progressive Relaxation Exercises — The trainer performed the PRE exercise online with the nurses. The video recording of the progressive relaxation exercises was shared with the nurses participating in the study on WhatsApp groups. Nurses were asked to perform the PRE application in accordance with the commands in the video recordings. In addition, a guide in which the steps of applying progressive relaxation exercises for each muscle group were written was given to the nurses. It was stated that they should do the application regularly for 25-30 minutes in the morning every day at home for a month. The PRE application was reminded daily from the WhatsApp group for the nurses to apply regularly to the sessions and not to disrupt the sessions. Nurses shared the messages stating that they were doing the PRE application on a daily basis for four weeks on WhatsApp groups.
  Arms: İntervention Group

SUMMARY:
This study was conducted to determine the effect of web-based progressive relaxation exercises applied to nurses working in a pandemic hospital on perceived stress and anxiety. In this randomized controlled clinical trial, nurses working in the pandemic hospital were randomly assigned to the control and intervention groups.

DETAILED DESCRIPTION:
The coronavirus disease-2019 (COVID-19) epidemic increases the stress and anxiety level of nurses due to many factors. This study was conducted to determine the effect of web-based progressive relaxation exercises applied to nurses working in a pandemic hospital on perceived stress and anxiety. In this randomized controlled clinical trial, nurses working in the pandemic hospital were randomly assigned to the control and intervention groups. The Web-Based Relaxation Exercises Program was trained and implemented online for 4 weeks by a trainer for the intervention group.The Perceived Stress Scale (PSS) and the State-Trait Anxiety Inventory (STAI) were completed online by participants in both groups before and after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-55
* Nurses working in the pandemic hospital

Exclusion Criteria:

* Nurses who did not agree to participate in the study
* Research Termination Criteria;
* Nurses who begin to receive support from a psychiatrist,
* Nurses who begin to use psychiatric medication,
* Nurses who are COVID positive,
* Moreover, the study was terminated with the nurses who wanted to leave the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Personal Information Form: | baseline
  Socio-demographic characteristics of nurses such as age, gender, educational status, working time in the profession, professional characteristics such as the unit they worked before and after the COVID-19 pandemic, working time and working style, how their family life was affected in the COVID-19 pandemic, and contains information on their greatest concern regarding the pandemic.
The Perceived Stress Scale | four weeks
  It is a five-point Likert-type scale and consists of 14 items. Participants rate each item on a scale ranging from "Never (0)" to "Very often (4)". Seven of the items with positive statements are scored in reverse. As the scores obtained from the scale increase, the perceived stress level of the person increases. PSS-14 scores range from 0 to 56, with 0-35 point range indicating normal stress level, 35-56 point range indicating that the individual is under stress.
State-Trait Anxiety Inventory | four weeks
  The 4-point Likert-type State Anxiety Inventory, consisting of 20 items in total, measures a person's anxiety at a certain time. According to the severity of the feelings, thoughts or behaviors expressed by the items in the State-Trait Anxiety Inventory, it is required to choose one of the options "not at all," "a little," "a lot," and "totally". There are 10 (items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20) reversed statements in the STAI. While scoring the scale, the reversed statements with a weight of 1 were converted to 4, and those with a weight of 4 were converted to 1. In direct statements, answers with a value of 4 indicate high anxiety. In reversed expressions, answers with a value of 1 indicate high anxiety, and a value of 4 indicates low anxiety. The last value obtained was accepted as the individual's anxiety score. It is reported that the level of anxiety is high for scores above 42 points.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagül Günaydın, Assist.Prof, Study Director — Yozgat Bozok University
Locations (1):
- Suleyman Demirel University, Merkez, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hersch RK, Cook RF, Deitz DK, Kaplan S, Hughes D, Friesen MA, Vezina M. Reducing nurses' stress: A randomized controlled trial of a web-based stress management program for nurses. Appl Nurs Res. 2016 Nov;32:18-25. doi: 10.1016/j.apnr.2016.04.003. Epub 2016 Apr 9. PMID 27969025
- [Background] Kackin O, Ciydem E, Aci OS, Kutlu FY. Experiences and psychosocial problems of nurses caring for patients diagnosed with COVID-19 in Turkey: A qualitative study. Int J Soc Psychiatry. 2021 Mar;67(2):158-167. doi: 10.1177/0020764020942788. Epub 2020 Jul 16. PMID 32674644
- [Background] Labrague LJ, De Los Santos JAA. COVID-19 anxiety among front-line nurses: Predictive role of organisational support, personal resilience and social support. J Nurs Manag. 2020 Oct;28(7):1653-1661. doi: 10.1111/jonm.13121. Epub 2020 Aug 21. PMID 32770780
- [Background] Hacimusalar Y, Kahve AC, Yasar AB, Aydin MS. Anxiety and hopelessness levels in COVID-19 pandemic: A comparative study of healthcare professionals and other community sample in Turkey. J Psychiatr Res. 2020 Oct;129:181-188. doi: 10.1016/j.jpsychires.2020.07.024. Epub 2020 Jul 21. PMID 32758711